CLINICAL TRIAL: NCT04463147
Title: Does the Needle-pilot Device Improve the Success of Vascular Catheterization Compared to the Classical Ultrasound-guided Technique
Acronym: NEEDLE-VISIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LOCAL/2019/AC-01
Record Dates: First submitted 2020-02-14; First posted 2020-07-09 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2021-08

CONDITIONS: Central Venous Catheters; Ultrasound Guidance
Keywords: Catheterization; Subclavian Vein; Vascular Access Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- new residents (Other): new residents in ultrasound-guided central vascular catheterization.
  Interventions: Device: Needle-pilotTM device
- experienced residents or ICU practitioners (Other): experienced residents or ICU practitioners in ultrasound-guided central vascular catheterization.
  Interventions: Device: Needle-pilotTM device

INTERVENTIONS:
Device: Needle-pilotTM device — The main objective aims to compare the procedure time between conventional real time ultrasound guidance and guidance with Needle-pilotTM device.

SUMMARY:
Real-time ultrasound guidance for central venous catheter catheterism is recommended in order to reduce complication, in particular for internal jugular site1. Nevertheless, the usefulness of ultrasound guidance for subclavian approach remains controversial, in particular because needle visualisation is more complex as compared to jugular site2,3. New magnetic devices (Needle-pilotTM device, Samsung Healthcare) could theoretically allow a better needle visualisation and a better success rate. The investigators hypothesize that such device could improve the feasibility of subclavian catheterism. As this device has not been evaluated in patients, the investigators decided to perform a simulation study on a human torso mannequin. This methodology has been already used by Vogel et al in 20154. The main objective aims to compare the procedure time between conventional real time ultrasound guidance and guidance with Needle-pilot™ device.

ELIGIBILITY:
Inclusion Criteria:

• all residents and practicioners of intensive care units in the Nîmes University Hospital, France.

Exclusion Criteria:

• unavailability or operator refusal, and more than one year without subclavian central catheterization (for experienced subgroup).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
First puncture success delay | during the procedure
  comparison of time (in seconds) between first puncture and successful "blood-aspiration" on a "subclavian venous" torso mannequin.

SECONDARY OUTCOMES:
Failure Rate | during the procedure
  Failure is defined as a puncture time > 300 seconds. The criterion corresponds to an absolute value: failure or not
Cutaneous wall | during the procedure
  Counting the number of times each participant will puncture the wall of the mannequin before succeeding in puncturing the vessel with the 2 techniques and comparing this number between groups.
Posterior wall | during the procedure
  Number of posterior vessel wall penetration
Puncture comfort | immediately after the procedure
  Operator puncture comfort feeling is assessed from 0 to 10 by each participants for each technique.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes, Hôpital Universitaire Carémeau, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grau-Mercier L, Chetioui A, Muller L, Roger C, Genre Grandpierre R, de La Coussaye JE, Cuvillon P, Claret PG, Bobbia X. Magnetic needle-tracking device for ultrasound guidance of radial artery puncture: A randomized study on a simulation model. J Clin Ultrasound. 2021 Mar;49(3):212-217. doi: 10.1002/jcu.22945. Epub 2020 Nov 16. PMID 33196110